CLINICAL TRIAL: NCT03766516
Title: A Multi-center and Non-interventional Registry of BrentuximabVedotinin Patients With Relapsed or Refractory Anaplastic Large Cell Lymphoma or Classical Hodgkin Lymphoma
Brief Title: Registry of BrentuximabVedotinin Patients With R/R Anaplastic Large Cell Lymphoma or Classical HL
Acronym: BRAVO
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Kim, Seok Jin, Principal Investigator, Samsung Medical Center
Other Study IDs: 2018-06-006
Record Dates: First submitted 2018-11-14; First posted 2018-12-06 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Relapsed or Refractory Anaplastic Large Cell Lymphoma & Hodgkin Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, Large-Cell, Anaplastic; Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: 1. Any patient planning to administer BrentuximabVedotin to treat the target disease.
  2. Any patient administering BrentuximabVedotin to treat the target disease.
  3. Any patient tracing BrentuximabVedotin after treating the target disease.
  4. Any patient administering another salvage option for cancer as the target disease has relapsed after terminating treatment using BrentuximabVedotin.

SUMMARY:
In case of relapsed or refractory ALK-negative ALCL patients, high-dosage chemotherapy/ stem cell transplantation is a universal salvage option for patients with sensitivity to anti-cancer treatment and a relatively successful salvage rate can be expected.

Recently, there has been a report of successful stem cell transplantation with full response to BrentuximabVedotin induced before stem cell transplantation and BrentuximabVedotin's role as a bridge therapy before stem cell transplantation has also been suggested.

Hodgkin lymphoma is a type of curable blood cancer with unique tissues and clinical characteristics. Based on the 2008 WHO classification, Hodgkin lymphoma has two types-nodular lymphocyte predominant type and classical type-and the classical type is further classified into four types, nodular sclerosis, mixed cellularity, lymphocyte depletion and lymphocyte-rich type.

Recently, immune checkpoint inhibitor is reported as a very effective treatment for relapsed Hodgkin lymphoma and more active treatment such as stem cell transplantation is considered for younger patients.

Treatment with Brentuximabvedotin targeting CD30+ is also very effective for the treatment of relapsed Hodgkin lymphoma and considered a good option for patients who are not suitable for stem cell transplantation or aged patients.

It shows consistent response to anti-CD30 antibody treatment in relation to relapsed anaplastic large cell lymphoma or Hodgkin lymphoma. The effect of Brentuximabvedotin (BV) has been proven for relapsed or intractable ALCL targeting CD30 as an antibody-chemical adhesive in the recent phase-2 study.

As Korea currently lacks real-world evidence in relation to BV, this study was conducted to address BV's effect as salvage therapy for patients with relapsed/refractoryanaplastic large cell lymphoma or Hodgkin lymphoma. This study identified the clinical results for treatment patterns and patients using the collected data and derived critical evidence for treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

Any patient subject to one of the following at the start of treatment with BrentuximabVedotin:

1. Any patient planning to administer BrentuximabVedotin to treat the target disease;
2. Any patient administering BrentuximabVedotin to treat the target disease;
3. Any patient tracing BrentuximabVedotin after treating the target disease; or
4. Any patient administering another salvage option for cancer as the target disease has relapsed after terminating treatment using BrentuximabVedotin.

Exclusion Criteria:

1. If conditions for target diseases are not met.
2. If conditions for target patients are not met.
3. If patients do not give written consent to participate in study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Any patient planning to administer BrentuximabVedotin to treat the target disease;
  2. Any patient administering BrentuximabVedotin to treat the target disease;
  3. Any patient tracing BrentuximabVedotin after treating the target disease; or
  4. Any patient administering another salvage option for cancer as the target disease has relapsed after terminating treatment using BrentuximabVedotin.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 3years
  Rate of patients with complete response and partial response based on Lugano classification.

SECONDARY OUTCOMES:
Response retention period | 3years
  From 1st dose date of Brentuximab Vedotin to progression date.
Overall survival period | 3years
  Period from start of salvage therapy with Brentuximab Vedotin to end of study.
Length of time until next treatment | 3years
  Length of time from start of salvage therapy with Brentuximab Vedotin to next salvage option after progress of disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No